CLINICAL TRIAL: NCT05442814
Title: Comparison of Anterior and Posterior Approaches of Suprascapular Nerve Block in Arthroscopic Shoulder Surgery
Brief Title: Anterior and Posterior Approaches of Suprascapular Nerve Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Ebru Girgin Dinç, MD, Principal Investigator, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EDinc
Record Dates: First submitted 2022-04-18; First posted 2022-07-05 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Shoulder Pain; Postoperative Pain; Diaphragmatic Paralysis; Subomohyoid Suprascapular Nerve Block; Anterior Suprascapular Nerve Block; Suprascapular Nerve Block
Keywords: Shoulder pain; Nerve Block; Diaphragmatic paralysis; Postoperative pain; Suprascapular block; Subomohyoid suprascapular block; Posterior Suprascapular block; Anterior Suprascapular block
MeSH Terms: conditions — Shoulder Pain; Pain, Postoperative; Respiratory Paralysis

STUDY DESIGN:
Intervention Model Description: participant with anterior suprascapular block ,group 1 participant with posterior suprascapular block, group 2
Who Masked: Outcomes Assessor
Masking Description: sealed envelope
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Posterior suprascapular block (Active Comparator): Suprascapular block performed by posterior approach
  Interventions: Procedure: Posterior suprascapular block
- Anterior suprascapular block (Active Comparator): Suprascapular block performed by anterior approach
  Interventions: Procedure: Anterior suprascapular block

INTERVENTIONS:
Procedure: Posterior suprascapular block — Diaphragmatic thickness fraction will be evaluated in the participant underwent suprascapular block performed by posterior approach
  Arms: Posterior suprascapular block
Procedure: Anterior suprascapular block — Diaphragmatic thickness fraction will be evaluated in the participant underwent suprascapular block performed by anterior approach
  Arms: Anterior suprascapular block

SUMMARY:
Suprascapular nerve is a mixed motor and sensory peripheral nerve arising from the superior trunk of brachial plexus.The suprascapular nerve runs through the posterior triangle of the neck, anterior of the trapezius muscle and dorsal of the omohyoid muscle, in direction of the scapula. Suprascapular nerve block is performed by anterior and posterior approach. Posterior approach of the suprascapular nerve block has been shown for many years to provide effective analgesia in the shoulder region for the chronic and acute pain. There are studies showing that suprascapular block with anterior approach provides effective analgesia in shoulder arthroscopy.

The aim of our study was to compare anterior and posterior approaches of suprascapular nerve block in terms of analgesic efficacy and patient safety.

DETAILED DESCRIPTION:
This study is a prospective randomized clinical trial will be conducted between March 2022 and March 2023.Participant will divide into two groups as participant who underwent suprascapular nerve block with the anterior approach and participant who underwent suprascapular nerve block with the posterior approach. Bupivacaine 5 ml %0.5 will be injected both group. Diaphragmatic thickness fraction will be evaluated with ultrasound left and right 7.-8. subcostal anterior axillary border with the participant with the semi-sitting position. Diaphragmatic thickness fraction will measure before the block and after 30 minutes the surgery. Participants will administered intravenous morphine patient controlled analgesia for 24 hours stay. The amount of opioid analgesics given in both groups will be determined (in mg). Postoperative 4th, 6th, 12th, 24th hour Visual Analogue Scale scores of the participants and opioid consumptions until that hours will be evaluated. An addition participant will be determined according to the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient who accepts to study protocol
* Scheduled for shoulder surgery
* Between the ages of 18 and 80

Exclusion Criteria:

* Patients with coagulopathy
* Patients with a history of local anesthetic drug allergy and toxicity
* Patients with advanced organ failure
* Patients with mental retardation
* Patients with infection present at the injection site
* Patients with diaphragm paralysis
* Pregnant patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Postoperative pain at the first postoperatively 30th. Min. | The first postoperative 30 minutes
  Visual analog scale (1-10): 1= no pain, 10= the worst pain ever feel.

SECONDARY OUTCOMES:
Diaphragmatic movements | Baseline (Before the block performed) and 30 minutes after the end of surgery
  Ratio of diaphragm thickness in end-inspiration and end-expiration measured by ultrasonography
Peroperatively opioid analgesic consumption (Remifentanil) | postoperative 0th.min
  milligram
Postoperative opioid analgesic consumption (morphine) | postoperative 30th. Min
  milligram
Postoperative opioid analgesic consumption (morphine) | postoperative 4 hours
  milligram
Postoperative opioid analgesic consumption (morphine) | postoperative 6 hours
  milligram
Postoperative opioid analgesic consumption (morphine) | postoperative 12 hours
  milligram
Postoperative opioid analgesic consumption (morphine) | postoperative 24 hours
  milligram
Postoperative pain at postoperative 4th. Hours | at postoperative 4th. Hours
  Visual analog scale (1-10): 1= no pain, 10= the worst pain ever feel.
Postoperative pain at postoperative 6th. Hours | at postoperative 6th. Hours
  Visual analog scale (1-10): 1= no pain, 10= the worst pain ever feel.
Postoperative pain at postoperative 12th. Hours | at postoperative 12th. Hours
  Visual analog scale (1-10): 1= no pain, 10= the worst pain ever feel.
Postoperative pain at postoperative 24th. Hours | at postoperative 24th. Hours
  Visual analog scale (1-10): 1= no pain, 10= the worst pain ever feel.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Girgin Dinç, MD, Principal Investigator — İstanbul Medeniyet University
Locations (1):
- Istanbul Medeniyet University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
After the article is accepted by the journal
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After the article is accepted by the journal
Access Criteria: After the article is accepted by the journal